CLINICAL TRIAL: NCT00084695
Title: The Use Of Umbilical Cord Blood As A Source Of Hematopoietic Stem Cells
Brief Title: Umbilical Cord Blood for Stem Cell Transplantation in Treating Young Patients With Malignant or Nonmalignant Diseases
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Kenneth Gerald Lucas, Penn State Children's Hospital
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000365544; PSCI-2003-232
Record Dates: First submitted 2004-06-10; First posted 2004-06-11 (Estimated); Last update posted 2014-01-10 (Estimated); Status verified 2008-10

CONDITIONS: Childhood Langerhans Cell Histiocytosis; Fanconi Anemia; Leukemia; Lymphoma; Myelodysplastic Syndromes; Neuroblastoma; Sarcoma; Unspecified Childhood Solid Tumor, Protocol Specific
Keywords: childhood myelodysplastic syndromes; recurrent childhood rhabdomyosarcoma; unspecified childhood solid tumor, protocol specific; previously treated childhood rhabdomyosarcoma; previously untreated childhood rhabdomyosarcoma; disseminated neuroblastoma; regional neuroblastoma; recurrent neuroblastoma; metastatic Ewing sarcoma/peripheral primitive neuroectodermal tumor; recurrent Ewing sarcoma/peripheral primitive neuroectodermal tumor; recurrent childhood acute lymphoblastic leukemia; juvenile myelomonocytic leukemia; childhood acute lymphoblastic leukemia in remission; childhood Burkitt lymphoma; recurrent childhood lymphoblastic lymphoma; stage III childhood lymphoblastic lymphoma; stage IV childhood lymphoblastic lymphoma; recurrent childhood small noncleaved cell lymphoma; stage III childhood small noncleaved cell lymphoma; stage IV childhood small noncleaved cell lymphoma; recurrent childhood large cell lymphoma; stage III childhood large cell lymphoma; stage IV childhood large cell lymphoma; stage III childhood Hodgkin lymphoma; stage IV childhood Hodgkin lymphoma; previously treated myelodysplastic syndromes; Fanconi anemia; de novo myelodysplastic syndromes; secondary myelodysplastic syndromes; childhood chronic myelogenous leukemia; chronic phase chronic myelogenous leukemia; relapsing chronic myelogenous leukemia; childhood Langerhans cell histiocytosis; recurrent childhood acute myeloid leukemia; recurrent/refractory childhood Hodgkin lymphoma
MeSH Terms: conditions — Fanconi Anemia; Leukemia; Lymphoma; Myelodysplastic Syndromes; Neuroblastoma; Sarcoma; Neuroectodermal Tumors, Primitive, Peripheral; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myelomonocytic, Juvenile; Burkitt Lymphoma; Dendritic Cell Sarcoma, Interdigitating; Leukemia, Myeloid, Chronic-Phase; Recurrence | interventions — Antilymphocyte Serum; Busulfan; Cyclophosphamide; fludarabine phosphate; Melphalan; Methylprednisolone; Radiotherapy

ARMS (4):
- Regimen A (Experimental): Patients undergo total body irradiation (TBI) two times daily on days -7 to -4. Patients receive cyclophosphamide IV over 30-60 minutes on days -3 and -2 and anti-thymocyte globulin (ATG) IV over at least 6 hours on days -3 to -1.
  Interventions: Biological: anti-thymocyte globulin; Drug: cyclophosphamide; Radiation: radiation therapy
- Regimen B (patients who do not receive TBI) (Experimental): Patients receive oral busulfan 4 times daily on days -8 to -5, and ATG IV over at least 6 hours and melphalan IV over 15-20 minutes on days -4 to -2.
  Interventions: Biological: anti-thymocyte globulin; Drug: busulfan; Drug: melphalan
- Regimen C (patients with Fanconi's anemia/related disorders) (Experimental): Patients undergo TBI on day -6. Patients receive ATG IV over at least 6 hours and methylprednisolone IV on days -5 to -1 and fludarabine IV over 30 minutes and cyclophosphamide IV over 30-60 minutes on days -5 to -2.
  Interventions: Biological: anti-thymocyte globulin; Drug: cyclophosphamide; Drug: fludarabine phosphate; Drug: methylprednisolone; Radiation: radiation therapy
- Regimen D (Experimental): Patients receive oral or IV busulfan 4 times daily on days -9 to -5, ATG IV over at least 6 hours on days -5 to -3, and cyclophosphamide IV over 30-60 minutes on days -5 to -2.
  Interventions: Biological: anti-thymocyte globulin; Drug: busulfan; Drug: cyclophosphamide

INTERVENTIONS:
Biological: anti-thymocyte globulin — Given IV
Drug: busulfan — Given orally
  Arms: Regimen B (patients who do not receive TBI); Regimen D
Drug: cyclophosphamide — Given IV
  Arms: Regimen A; Regimen C (patients with Fanconi's anemia/related disorders); Regimen D
Drug: fludarabine phosphate — Given IV
  Arms: Regimen C (patients with Fanconi's anemia/related disorders)
Drug: melphalan — Given IV
  Arms: Regimen B (patients who do not receive TBI)
Drug: methylprednisolone — Given IV
  Arms: Regimen C (patients with Fanconi's anemia/related disorders)
Radiation: radiation therapy — Patients undergo radiation therapy two times daily on days -7 to -4.
  Arms: Regimen A; Regimen C (patients with Fanconi's anemia/related disorders)

SUMMARY:
RATIONALE: Umbilical cord blood transplantation may be able to replace immune cells that were destroyed by chemotherapy or radiation therapy.

PURPOSE: This phase II trial is studying how well umbilical cord blood works as a source of stem cells in treating patients with types of cancer as well as other diseases.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the impact of the use of umbilical cord blood as a source of hematopoietic stem cells for children with life-threatening oncologic, hematologic, or genetic/metabolic disorders in need of a stem cell transplant.
* Compare the incidence of graft-versus-host disease in patients receiving cord blood transplants in this study with historical data for unrelated donor stem cell transplants.
* Compare the incidence of engraftment in patients receiving cord blood transplants in this study with historical data for unrelated donor stem cell transplants.

OUTLINE:

* Preparative therapy: Patients are treated on 1 of 4 preparative therapy regimens.

  * Regimen A: Patients undergo total body irradiation (TBI) two times daily on days -7 to -4. Patients receive cyclophosphamide IV over 30-60 minutes on days -3 and -2 and anti-thymocyte globulin (ATG) IV over at least 6 hours on days -3 to -1.
  * Regimen B (patients who do not receive TBI): Patients receive oral busulfan 4 times daily on days -8 to -5, and ATG IV over at least 6 hours and melphalan IV over 15-20 minutes on days -4 to -2.
  * Regimen C (patients with Fanconi's anemia and related disorders): Patients undergo TBI on day -6. Patients receive ATG IV over at least 6 hours and methylprednisolone IV on days -5 to -1 and fludarabine IV over 30 minutes and cyclophosphamide IV over 30-60 minutes on days -5 to -2.
  * Regimen D: Patients receive oral or IV busulfan 4 times daily on days -9 to -5, ATG IV over at least 6 hours on days -5 to -3, and cyclophosphamide IV over 30-60 minutes on days -5 to -2.
* Cord blood transplant: All patients undergo umbilical cord blood transplantation on day 0.
* Graft-versus-host disease prophylaxis: Patients receive oral or IV cyclosporine twice daily beginning on day -1. Patients also receive methylprednisolone IV twice daily beginning on day 5 and continuing until at least day 28.

PROJECTED ACCRUAL: A total of 25 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of malignant or non-malignant disease, including but not limited to any of the following:

  * Acute myeloid leukemia or acute lymphoblastic leukemia (ALL) with resistant disease beyond first clinical remission (CR)
  * ALL in first CR at high-risk because of 1 of the following factors:

    * Hypoploidy
    * Pseudodiploidy with translocations t(9;22), t(4;11), or t(8;14)
    * Elevated WBC at diagnosis as follows:

      * > 100,000/mm^3 for patients 6-12 months of age
      * > 50,000/mm^3 for patients 10-20 years of age
      * > 20,000/mm^3 for patients 21 years of age
    * Burkitt's lymphoma/leukemia
  * Chronic myelogenous leukemia in first chronic phase or beyond
  * Juvenile myelomonocytic leukemia
  * Advanced stage or relapsed lymphoma
  * Advanced stage or relapsed solid tumors, including any of the following:

    * Neuroblastoma
    * Ewing's sarcoma
    * Rhabdomyosarcoma
  * Myelodysplastic syndromes, excluding patients with grade 3 or 4 myelofibrosis
  * Familial erythrophagocytic histiocytosis
  * Histiocytosis unresponsive to medical management
  * Inborn errors of metabolism
  * Langerhans cell histiocytosis unresponsive to medical management
  * Immune deficiencies, including:

    * Severe combined immune deficiency
    * Wiskott-Aldrich
  * Hemoglobinopathies, including sickle cell disease and thalassemia
  * Severe aplastic anemia
  * Fanconi's anemia
  * Metabolic storage diseases
* Unrelated cord blood donor must be HLA-identical OR may be mismatched for 1, 2, or 3 HLA-loci (A, B, DR)
* No other existing HLA-identical related donor available at the time of transplantation

PATIENT CHARACTERISTICS:

Age

* 21 and under

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* See Disease Characteristics

Hepatic

* Not specified

Renal

* Not specified

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 25 (Estimated)
Dates: Start 2003-09; Primary Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Impact of the use of umbilical cord blood as a source of hematopoietic stem cells
Comparison of the incidence of graft-vs-host disease with historical data
Comparison of the incidence of engraftment with historical data

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth G. Lucas, MD, Study Chair — Milton S. Hershey Medical Center
Locations (1):
- Penn State Hershey Cancer Institute at Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States